CLINICAL TRIAL: NCT03023813
Title: Individualizing Disease Prevention for Middle-Aged Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated on 2/17/2021 due to on-going and uncertain nature of COVID-19 pandemic; this was not a suspension of IRB approval.
Sponsor: Glen Taksler (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Glen Taksler, Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-854
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Primary Health Care
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Multiple round pilot testing. Some round(s) will have a single group with 1 arm. Other round(s) will be parallel with 2 arms.
Masking Description: Only the 2 arm round(s) will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Individualized preventive care recommendations will be distributed to subjects.
  Interventions: Other: Intervention
- Control (No Intervention): Usual care
- Development Phase (Experimental): Non-randomized receipt of individualized preventive care recommendations
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Written material provided.
  Arms: Development Phase; Intervention

SUMMARY:
The primary objective of this study is to help patients compare the benefits of various preventive care services, based on their individual risk factors (such as smoking status, obesity, high blood pressure, high cholesterol, etc.). A tailored decision tool will be provided to each participant during primary care appointments to facilitate discussion between the participant and his/her provider regarding prioritizing preventive service recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an appointment with primary care provider during study period
* Two or more of the following risk factors:
* Tobacco use
* Overweight/obese
* Hypertension
* Hyperlipidemia
* Diabetes
* Alcohol Misuse
* Depression
* History of Sexually Transmitted Infection
* Being overdue for the following screenings: Colorectal, cervical, breast, lung

Exclusion Criteria:

- Severely limited life expectancy (cancer, congestive heart failure, chronic obstructive pulmonary disease, end stage renal disease)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen Taksler, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krist AH, Glenn BA, Glasgow RE, Balasubramanian BA, Chambers DA, Fernandez ME, Heurtin-Roberts S, Kessler R, Ory MG, Phillips SM, Ritzwoller DP, Roby DH, Rodriguez HP, Sabo RT, Sheinfeld Gorin SN, Stange KC; MOHR Study Group. Designing a valid randomized pragmatic primary care implementation trial: the my own health report (MOHR) project. Implement Sci. 2013 Jun 25;8:73. doi: 10.1186/1748-5908-8-73. PMID 23799943
- [Background] Glasgow RE, Kessler RS, Ory MG, Roby D, Gorin SS, Krist A. Conducting rapid, relevant research: lessons learned from the My Own Health Report project. Am J Prev Med. 2014 Aug;47(2):212-9. doi: 10.1016/j.amepre.2014.03.007. Epub 2014 Jun 18. PMID 24953520
- [Background] Edwards A, Elwyn G. Inside the black box of shared decision making: distinguishing between the process of involvement and who makes the decision. Health Expect. 2006 Dec;9(4):307-20. doi: 10.1111/j.1369-7625.2006.00401.x. PMID 17083558
- [Background] Elwyn G, Edwards A, Wensing M, Hood K, Atwell C, Grol R. Shared decision making: developing the OPTION scale for measuring patient involvement. Qual Saf Health Care. 2003 Apr;12(2):93-9. doi: 10.1136/qhc.12.2.93. PMID 12679504
- [Background] Nagykaldi Z, Aspy CB, Chou A, Mold JW. Impact of a Wellness Portal on the delivery of patient-centered preventive care. J Am Board Fam Med. 2012 Mar-Apr;25(2):158-67. doi: 10.3122/jabfm.2012.02.110130. PMID 22403196
- [Background] Sepucha KR, Fagerlin A, Couper MP, Levin CA, Singer E, Zikmund-Fisher BJ. How does feeling informed relate to being informed? The DECISIONS survey. Med Decis Making. 2010 Sep-Oct;30(5 Suppl):77S-84S. doi: 10.1177/0272989X10379647. PMID 20881156
- [Background] Dillard AJ, Ferrer RA, Ubel PA, Fagerlin A. Risk perception measures' associations with behavior intentions, affect, and cognition following colon cancer screening messages. Health Psychol. 2012 Jan;31(1):106-13. doi: 10.1037/a0024787. Epub 2011 Aug 1. PMID 21806302
- [Background] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Phillips SM, Glasgow RE, Bello G, Ory MG, Glenn BA, Sheinfeld-Gorin SN, Sabo RT, Heurtin-Roberts S, Johnson SB, Krist AH; MOHR Study Group. Frequency and prioritization of patient health risks from a structured health risk assessment. Ann Fam Med. 2014 Nov-Dec;12(6):505-13. doi: 10.1370/afm.1717. PMID 25384812
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Fagerlin A, Zikmund-Fisher BJ, Ubel PA, Jankovic A, Derry HA, Smith DM. Measuring numeracy without a math test: development of the Subjective Numeracy Scale. Med Decis Making. 2007 Sep-Oct;27(5):672-80. doi: 10.1177/0272989X07304449. Epub 2007 Jul 19. PMID 17641137
- [Background] Zikmund-Fisher BJ, Smith DM, Ubel PA, Fagerlin A. Validation of the Subjective Numeracy Scale: effects of low numeracy on comprehension of risk communications and utility elicitations. Med Decis Making. 2007 Sep-Oct;27(5):663-71. doi: 10.1177/0272989X07303824. Epub 2007 Jul 24. PMID 17652180
- [Background] Tait AR, Voepel-Lewis T, Zikmund-Fisher BJ, Fagerlin A. Presenting research risks and benefits to parents: does format matter? Anesth Analg. 2010 Sep;111(3):718-23. doi: 10.1213/ANE.0b013e3181e8570a. Epub 2010 Aug 4. PMID 20686011
- [Background] Tait AR, Zikmund-Fisher BJ, Fagerlin A, Voepel-Lewis T. Effect of various risk/benefit trade-offs on parents' understanding of a pediatric research study. Pediatrics. 2010 Jun;125(6):e1475-82. doi: 10.1542/peds.2009-1796. Epub 2010 May 10. PMID 20457688
- [Background] Hawley ST, Zikmund-Fisher B, Ubel P, Jancovic A, Lucas T, Fagerlin A. The impact of the format of graphical presentation on health-related knowledge and treatment choices. Patient Educ Couns. 2008 Dec;73(3):448-55. doi: 10.1016/j.pec.2008.07.023. Epub 2008 Aug 27. PMID 18755566
- [Background] Tait AR, Voepel-Lewis T, Zikmund-Fisher BJ, Fagerlin A. The effect of format on parents' understanding of the risks and benefits of clinical research: a comparison between text, tables, and graphics. J Health Commun. 2010 Jul;15(5):487-501. doi: 10.1080/10810730.2010.492560. PMID 20677054
- [Background] Lloyd A, Joseph-Williams N, Edwards A, Rix A, Elwyn G. Patchy 'coherence': using normalization process theory to evaluate a multi-faceted shared decision making implementation program (MAGIC). Implement Sci. 2013 Sep 5;8:102. doi: 10.1186/1748-5908-8-102. PMID 24006959
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Derived] Taksler GB, Hu B, DeGrandis F Jr, Montori VM, Fagerlin A, Nagykaldi Z, Rothberg MB. Effect of Individualized Preventive Care Recommendations vs Usual Care on Patient Interest and Use of Recommendations: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2131455. doi: 10.1001/jamanetworkopen.2021.31455. PMID 34726747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control | Development Phase
Started | 39 | 34 | 31
Completed | 38 | 32 | 31
Not Completed | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Development Phase | Total
Number analyzed (Participants) | 38 | 32 | 31 | 101
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 55.9 [53 to 59] | 56.6 [53 to 61] | 56.9 [53 to 61] | 56.5 [53 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 23 | 73
  Male | 13 | 7 | 8 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 1 | 4
  Black or African American | 30 | 22 | 28 | 80
  White | 5 | 10 | 2 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 32 | 31 | 101
Practice site [Count of Participants; unit: Participants] — Study was conducted at 3 physical locations (primary care ambulatory clinics), denoted as Site 1, Site 2 or Site 3.
  Participants
    Site 1 | 20 | 17 | 14 | 51
    Site 2 | 14 | 12 | 17 | 43
    Site 3 | 4 | 3 | 0 | 7
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 4 | 1 | 6
  High school (diploma or GED) | 12 | 6 | 14 | 32
  Some college | 13 | 6 | 10 | 29
  College degree | 3 | 9 | 5 | 17
  Masters degree | 5 | 3 | 0 | 8
  Doctoral or professional degree | 0 | 0 | 1 | 1
  Missing | 4 | 4 | 0 | 8
Marital status [Count of Participants; unit: Participants]
  Married or civil/domestic partner | 14 | 12 | 8 | 34
  Widowed | 2 | 4 | 3 | 9
  Divorced | 7 | 3 | 9 | 19
  Separated | 3 | 3 | 2 | 8
  Never married | 12 | 10 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Interest in Individualized Preventive Care Recommendations.
Description: Measured by individualized preventive service recommendations, tailored to patient's specific medical conditions. Measured by surveys.
  Survey question: "Overall, how helpful did you find the written materials (handouts)?" Ten point scale (minimum 1, maximum 10, higher score is better outcome)
Time Frame: Within 3 days of index primary care appointment.
Population: Patients who completed surveys
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
score on a scale | 8.9 [8 to 10] | NA [NA to NA] — Collected from intervention subjects only | 9.0 [8 to 10]

2. Primary Outcome: Interest in Individualized Preventive Care Recommendations.
Description: Measured by individualized preventive service recommendations, tailored to patient's specific medical conditions. Measured by surveys.
  Survey question: "In the future, would you like to see updated written materials (handouts)?" Ten point scale (minimum 1, maximum 10, higher score is better outcome)
Time Frame: Within 3 days of index primary care appointment.
Population: Patients who completed surveys
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
score on a scale | 9.0 [9 to 10] | NA [NA to NA] — Collected from intervention subjects only | 9.0 [9 to 10]

3. Secondary Outcome: Use of Shared Decision Making.
Description: Measured by surveys. Survey metric: Shared Decision Making (SDM)-Q-9 validated scale, converted to 100 point denominator 100 point scale (minimum 1, maximum 100, higher score is better outcome)
Time Frame: Within 3 days of index primary care appointment.
Population: Patients who completed surveys
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
score on a scale | 79.0 (4.6) | 74.3 (5.1) | 86.4 (2.6)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = 0.50, t-test, 2 sided

4. Secondary Outcome: Patient Readiness to Change Health Behaviors.
Description: Measured by surveys. Proportion of top-3 individualized preventive service recommendations ready to change over next 1 month Numerator: Number of top-3-ranked recommendations with score >=6 out of 7 on Likert scale for readiness to change over next 1 month (minimum=1, maximum=7, higher score was better) Denominator: The number of individualized preventive service recommendations provided to a patient or 3, whichever was lower
Time Frame: Within 3 days of index primary care appointment.
Population: Patients who completed surveys
Measure: Mean (Standard Error); unit: percentage of survey responses
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
percentage of survey responses | 84.6 (7.2) | 70.8 (9.5) | 83.3 (6.9)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .25, t-test, 2 sided

5. Secondary Outcome: Patient Readiness to Change Health Behaviors
Description: Measured by surveys Proportion of top-3 individualized preventive service recommendations ready to change over next 2-6 months Numerator: Number of top-3-ranked recommendations with score >=6 out of 7 on Likert scale for readiness to change over next 2-6 months (minimum=1, maximum=7, higher score was better) Denominator: The number of individualized preventive service recommendations provided to a patient or 3, whichever was lower
Time Frame: Within 3 days of index primary care appointment
Population: Patients who completed surveys
Measure: Mean (Standard Error); unit: percentage of survey responses
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
percentage of survey responses | 83.3 (7.8) | 72.7 (9.7) | 86.7 (6.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = .39, t-test, 2 sided

6. Secondary Outcome: Patient Readiness to Change Health Behaviors.
Description: Measured by surveys Proportion of bottom-3 individualized preventive service recommendations ready to change over next 1 month Numerator: Number of bottom-3-ranked recommendations with score >=6 out of 7 on Likert scale for readiness to change over next 1 month (minimum=1, maximum=7, higher score was better) Denominator: The number of individualized preventive service recommendations provided to a patient or 3, whichever was lower
Time Frame: Within 3 days of index primary care appointment
Population: Patients who completed surveys
Measure: Mean (Standard Error); unit: percentage of survey responses
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
percentage of survey responses | 70.4 (9.0) | 77.8 (10.1) | 78.6 (7.9)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = 0.59, t-test, 2 sided

7. Secondary Outcome: Patient Readiness to Change Health Behaviors
Description: Measured by surveys. Proportion of bottom-3 individualized preventive service recommendations ready to change over next 2-6 months Numerator: Number of bottom-3-ranked recommendations with score >=6 out of 7 on Likert scale for readiness to change over next 2-6 months (minimum=1, maximum=7, higher score was better) Denominator: The number of individualized preventive service recommendations provided to a patient or 3, whichever was lower
Time Frame: Within 3 days of index primary care appointment
Population: Patients who completed surveys
Measure: Mean (Standard Error); unit: percentage of survey responses
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 31
percentage of survey responses | 80.0 (10.7) | 69.2 (13.3) | 82.1 (7.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = 0.53, t-test, 2 sided

8. Secondary Outcome: Decisional Comfort.
Description: Measured by surveys. Survey metric: Decisional Conflict Scale (validated scale), converted to 100 point denominator 100 point scale (minimum 1, maximum 100, higher score is better outcome)
Time Frame: Within 3 days of index primary care appointment.
Population: Patients who completed surveys (Data not collected for Development Phase)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 0
score on a scale | 73.2 (5.3) | 72.3 (5.8) |
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; p = 0.91, t-test, 2 sided

9. Secondary Outcome: Preventive Care Outcomes for Patients.
Description: Number of participants with at least 1 follow-up encounter during the 1 year after an index encounter.
Time Frame: Within 1 year of index primary care appointment.
Population: Outcome tables are not included for specific preventive services because outcomes were not assessed by arm (instead, a statistical regression strategy was used).
  This outcome was not collected for participants in the Development arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control | Development Phase
Number analyzed (Participants) | 38 | 32 | 0
Participants | 31 | 30 | 0
Statistical Analysis 1: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included weight loss; Test type: Other — Percent change in weight (lbs.) since the baseline encounter; p = 0.27, Mixed Models Analysis; Mean Difference (Net) = -2.96, 95% CI 2-sided [-8.18 to 2.26] — Result for intervention arm minus control arm
Statistical Analysis 2: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included blood pressure control; Test type: Other — Change in systolic blood pressure since the baseline encounter (mmHg); p = 0.19, Mixed Models Analysis; Mean Difference (Net) = -6.42, 95% CI 2-sided [-16.12 to 3.27] — Result for intervention arm minus control arm
Statistical Analysis 3: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included glycemic control; Test type: Other — Percentage point change in HbA1c (%) since the baseline encounter; p = 0.24, Mixed Models Analysis; Mean Difference (Net) = -0.68, 95% CI 2-sided [-1.82 to 0.45] — Result for intervention arm minus control arm
Statistical Analysis 4: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included lipids control; Test type: Other — Percentage point change in 10-year atherosclerotic cardiovascular disease risk (%), as estimated by the American College of Cardiology Pooled Cohort Equations, since the baseline encounter; p = 0.34, Generalized linear mixed regression; Mean Difference (Net) = -1.20, 95% CI 2-sided [-3.65 to 1.26] — Result for intervention arm minus control arm
Statistical Analysis 5: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included lipids control; Test type: Other — Change in low-density lipoprotein (LDL) cholesterol (mg/dL) since the baseline encounter; p = 0.36, Mixed Models Analysis; Mean Difference (Net) = -8.46, 95% CI 2-sided [-26.63 to 9.70] — Result for intervention arm minus control arm
Statistical Analysis 6: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included tobacco cessation; Test type: Other — Change in smoking intensity (defined as a change in smoking status from Current Every Day to either Current Some Days or Quit; or from Current Some Days to Quit) since the baseline encounter; p = 0.92, Mixed Models Analysis; Generalized linear mixed regression with logit link; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.03 to 45.56] — Result for intervention arm relative to control arm. OR <1 indicates reduction in smoking intensity; OR >1 indicates increase in smoking intensity
Statistical Analysis 7: Comparison: Intervention vs Control; Among participants whose individualized preventive care recommendations included colorectal cancer screening; Test type: Other — Receipt of colorectal cancer screening since the baseline encounter; p = 0.99, Mixed Models Analysis; Generalized linear mixed regression with logit link; Odds Ratio (OR) = 2.52, 95% CI 2-sided [0.001 to 1000] — Result for intervention arm relative to control arm. Lower limit estimate was <0.001 and upper limit estimate was >1000 (ClinicalTrials.gov does not allow < or > to be entered into the confidence interval lower limit or upper limit fields)

ADVERSE EVENTS:
Time Frame: Up to 1 year following enrollment of each patient participant.
Description: As an Institutional Review Board (IRB)-determined minimal risk study, adverse events were not tracked by the study team. Instead, participants were asked to report any adverse events to the study team or the IRB. No events were reported.
Arm/Group | Intervention | Control | Development Phase
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/38 | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03023813/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03023813/ICF_001.pdf